CLINICAL TRIAL: NCT00996918
Title: A Phase 3 Extension, Multicenter, Double-Blind, Long-Term Safety And Tolerability Trial Of Bapineuzumab (AAB-001, ELN115727) In Subjects With Alzheimer Disease Who Are Apolipoprotein E e4 Noncarriers And Participated In Study 3133K1-3000
Brief Title: A Long-Term Safety And Tolerability Study Of Bapineuzumab In Alzheimer Disease Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated on August 6, 2012, because 2 large Phase 3 studies showed no clinical benefit. This decision was not based on any new safety concerns.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3133K1-3002; B2521003
Record Dates: First submitted 2009-10-14; First posted 2009-10-16 (Estimated); Results first posted 2014-01-01 (Estimated); Last update posted 2014-01-01 (Estimated); Status verified 2013-11

CONDITIONS: Alzheimer Disease
Keywords: antibody
MeSH Terms: conditions — Alzheimer Disease | interventions — bapineuzumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bapineuzumab 0.5 mg/kg (Experimental): bapineuzumab
  Interventions: Drug: Bapineuzumab 0.5 mg/kg
- Bapineuzumab 1.0 m/kg (Experimental): bapineuzumab
  Interventions: Drug: Bapineuzumab 1.0 m/kg

INTERVENTIONS:
Drug: Bapineuzumab 0.5 mg/kg — Bapineuzumab I.V., 0.5 mg/kg, infusion every 13 weeks for a total of 16 infusions.
  Other Names: AAB-001
  Arms: Bapineuzumab 0.5 mg/kg
Drug: Bapineuzumab 1.0 m/kg — I.V., 1.0 mg/kg, infusion every 13 weeks for a total of 16 infusions.
  Other Names: AAB-001
  Arms: Bapineuzumab 1.0 m/kg

SUMMARY:
The purpose of this study is to assess the long-term safety and tolerability of bapineuzumab in subjects with Alzheimer Disease who participated in study 3133K1-3000 (NCT00667810). Over 250 sites will participate in over 26 countries. Subjects will receive bapineuzumab. Each subject's participation will last approximately 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Subject has completed study 3133K1-3000 and brain magnetic resonance imaging (MRI) scan consistent with the diagnosis of Alzheimer Disease
* Mini-Mental Status Examination (MMSE) >=10 at screening
* Caregiver able to attend all clinic visits with subject

Exclusion Criteria:

* Any medical or psychiatric contraindication or clinically significant abnormality that, in the investigator's judgment, will substantially increase the risk associated with the subject's participation in and completion of the study or could preclude the evaluation of the subject's response.
* Any significant brain MRI abnormality.
* Use of any investigational drugs or devices, other than bapineuzumab within the last 60 days prior to screening

Min Age: 51 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2009-12; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (71):
- Australia (5):
  - Pfizer Investigational Site, Hornsby, New South Wales
  - Pfizer Investigational Site, Adelaide, South Australia
  - Pfizer Investigational Site, Woodville South, South Australia
  - Pfizer Investigational Site, Heidelberg Heights, Victoria
  - Pfizer Investigational Site, Nedlands, Western Australia
- Belgium (3):
  - Pfizer Investigational Site, Antwerp
  - Pfizer Investigational Site, Brussels
  - Pfizer Investigational Site, Edegem
- Pfizer Investigational Site, Santiago, Chile, Chile
- Finland (2):
  - Pfizer Investigational Site, Kuopio
  - Pfizer Investigational Site, Turku
- France (13):
  - Pfizer Investigational Site, Dijon, France
  - Pfizer Investigational Site, Lille, France
  - Pfizer Investigational Site, Marseille, France
  - Pfizer Investigational Site, Paris, France
  - Pfizer Investigational Site, Caen
  - Pfizer Investigational Site, Marseille
  - Pfizer Investigational Site, Montpellier
  - Pfizer Investigational Site, Nantes - Saint Herblain
  - Pfizer Investigational Site, Nice
  - Pfizer Investigational Site, Poitiers
  - Pfizer Investigational Site, Rennes
  - Pfizer Investigational Site, Rouen
  - Pfizer Investigational Site, Toulouse
- Italy (2):
  - Pfizer Investigational Site, Milan
  - Pfizer Investigational Site, Roma
- Japan (13):
  - Pfizer Investigational Site, Aichi
  - Pfizer Investigational Site, Chiba
  - Pfizer Investigational Site, Fukuoka
  - Pfizer Investigational Site, Hiroshima
  - Pfizer Investigational Site, Hyōgo
  - Pfizer Investigational Site, Kagawa
  - Pfizer Investigational Site, Kanagawa
  - Pfizer Investigational Site, Kyoto
  - Pfizer Investigational Site, Nagano
  - Pfizer Investigational Site, Okayama
  - Pfizer Investigational Site, Osaka
  - Pfizer Investigational Site, Shizuoka
  - Pfizer Investigational Site, Tokyo
- Netherlands (2):
  - Pfizer Investigational Site, 's-Hertogenbosch
  - Pfizer Investigational Site, Leeuwarden
- Pfizer Investigational Site, North Shore, NZ, New Zealand
- Poland (4):
  - Pfizer Investigational Site, Poznan, Poland
  - Pfizer Investigational Site, Bydgoszcz
  - Pfizer Investigational Site, Krakow
  - Pfizer Investigational Site, Warsaw
- Portugal (3):
  - Pfizer Investigational Site, Amadora, Amadora
  - Pfizer Investigational Site, Coimbra, Coimbra District
  - Pfizer Investigational Site, Lisbon, Lisbon District
- Slovakia (2):
  - Pfizer Investigational Site, Bratislava
  - Pfizer Investigational Site, Rimavská Sobota
- South Africa (2):
  - Pfizer Investigational Site, Johannesburg, Gauteng
  - Pfizer Investigational Site, Pretoria, Gauteng
- Spain (8):
  - Pfizer Investigational Site, Elche, Alicante
  - Pfizer Investigational Site, Palma de Mallorca, Balearic Islands
  - Pfizer Investigational Site, Barcelona, Barcelona
  - Pfizer Investigational Site, Terrassa, Barcelona
  - Pfizer Investigational Site, Burgos, Burgos
  - Pfizer Investigational Site, Plasencia, Caceres
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, Madrid
- Pfizer Investigational Site, Malmo, Sweden
- Pfizer Investigational Site, Basel, Canton of Basel-City, Switzerland
- United Kingdom (8):
  - Pfizer Investigational Site, London, London
  - Pfizer Investigational Site, Brighton
  - Pfizer Investigational Site, Glasgow
  - Pfizer Investigational Site, London
  - Pfizer Investigational Site, Newcastle upon Tyne
  - Pfizer Investigational Site, Penarth
  - Pfizer Investigational Site, Sheffield
  - Pfizer Investigational Site, Swindon

REFERENCES:
- [Derived] Ivanoiu A, Pariente J, Booth K, Lobello K, Luscan G, Hua L, Lucas P, Styren S, Yang L, Li D, Black RS, Brashear HR, McRae T. Long-term safety and tolerability of bapineuzumab in patients with Alzheimer's disease in two phase 3 extension studies. Alzheimers Res Ther. 2016 Jun 23;8(1):24. doi: 10.1186/s13195-016-0193-y. PMID 27334799
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3133K1-3002&StudyName=A%20Long-Term%20Safety%20And%20Tolerability%20Study%20Of%20Bapineuzumab%20In%20Alzheimer%20Disease%20Patients

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This extension study was conducted at 91 centers in 17 countries. The study was terminated early by the sponsor on 06 August 2012. Participants who had not completed the final follow-up visit prior to 06 August 2012 were asked to complete an early termination visit.
Pre-assignment Details: Participants who had completed the base study protocol 3133K1-3000 were allowed to participate in this extension study. Participants who developed vasogenic edema during study 3133K1-3000 were considered for study 3133K1-3002 participation if the abnormality was resolved and the participant met criteria to resume the investigational product.
Groups:
- Placebo/Bapineuzumab 0.5 Milligram/Kilogram(mg/kg): Participants received placebo in the base study and 0.5 mg/kg bapineuzumab in this extension study. In this extension study bapineuzumab was administered by IV infusion approximately every 13 weeks up to Week 195.
- Bapineuzumab 0.5 mg/kg/ Bapineuzumab 0.5 mg/kg: Participants received 0.5 mg/kg bapineuzumab in both the base and extension studies. In this extension study bapineuzumab was administered by IV infusion approximately every 13 weeks up to Week 195.
- Placebo/Bapineuzumab 1.0 mg/kg: Participants received placebo in the base study and 1.0 mg/kg bapineuzumab in this extension study. In this extension study bapineuzumab was administered by IV infusion approximately every 13 weeks up to Week 195.
- Bapineuzumab 1.0 mg/kg/Bapineuzumab 1.0 mg/kg: Participants received 1.0 mg/kg bapineuzumab in both the base and extension studies. In this extension study bapineuzumab was administered by IV infusion approximately every 13 weeks up to Week 195.
- Bapineuzumab 2.0 mg/kg/ Bapineuzumab 1.0 mg/kg: Participants originally randomized to 2.0 mg/kg bapineuzumab were reassigned to the 1.0 mg/kg dose level after discontinuation of 2.0 mg/kg dose level in the base study and continued the 1.0 mg/kg dose in this extension study. In this extension study bapineuzumab was administered by IV infusion approximately every 13 weeks up to Week 195.
Period: Overall Study
Arm/Group | Placebo/Bapineuzumab 0.5 Milligram/Kilogram(mg/kg) | Bapineuzumab 0.5 mg/kg/ Bapineuzumab 0.5 mg/kg | Placebo/Bapineuzumab 1.0 mg/kg | Bapineuzumab 1.0 mg/kg/Bapineuzumab 1.0 mg/kg | Bapineuzumab 2.0 mg/kg/ Bapineuzumab 1.0 mg/kg
Started | 39 | 66 | 37 | 56 | 4
Treated | 39 | 66 | 37 | 56 | 4
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 39 | 66 | 37 | 56 | 4
Not completed — Lack of Efficacy | 1 | 1 | 2 | 2 | 0
Not completed — Adverse Event | 2 | 5 | 2 | 6 | 0
Not completed — Withdrawal by Subject | 1 | 4 | 3 | 3 | 2
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0
Not completed — Discontinuation of Study by Sponsor | 31 | 54 | 30 | 45 | 2
Not completed — Loss of Caregiver | 0 | 1 | 0 | 0 | 0
Not completed — Other | 3 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo/Bapineuzumab 0.5 mg/kg: Participants received placebo in the base study and 0.5 mg/kg bapineuzumab in this extension study. In this extension study bapineuzumab was administered by IV infusion approximately every 13 weeks up to Week 195.
- Bapineuzumab 2.0 mg/kg/Bapineuzumab 1.0 mg/kg: Participants originally randomized to 2.0 mg/kg bapineuzumab were reassigned to the 1.0 mg/kg dose level after discontinuation of 2.0 mg/kg dose level in the base study and continued the 1.0 mg/kg dose in this extension study. In this extension study bapineuzumab was administered by IV infusion approximately every 13 weeks up to Week 195.
- Total: Total of all reporting groups
Arm/Group | Placebo/Bapineuzumab 0.5 mg/kg | Bapineuzumab 0.5 mg/kg/ Bapineuzumab 0.5 mg/kg | Placebo/Bapineuzumab 1.0 mg/kg | Bapineuzumab 1.0 mg/kg/Bapineuzumab 1.0 mg/kg | Bapineuzumab 2.0 mg/kg/Bapineuzumab 1.0 mg/kg | Total
Number analyzed (Participants) | 38 | 62 | 33 | 53 | 4 | 190
Age Continuous [Mean (Standard Deviation); unit: Years] | 68.9 (9.70) | 71.9 (8.83) | 68.8 (8.59) | 70.6 (9.13) | 71.3 (10.63) | 70.4 (9.08)
Age, Customized [Number; unit: Number of participants]
  < 65 | 17 | 15 | 12 | 17 | 1 | 62
  >= 65 | 21 | 47 | 21 | 36 | 3 | 128
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 28 | 14 | 19 | 3 | 77
  Male | 25 | 34 | 19 | 34 | 1 | 113

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting a Serious Adverse Event.
Description: Safety was measured according to standard adverse event collection as described in the Adverse Event Section of the Results. Complete tables of events are provided there.
Time Frame: Up to Week 195
Population: The Safety Population included all participants who consented to participate in the extension and received at least one dose of the investigational product (in the extension study).
Measure: Number; unit: Number of participants
Arm/Group | Placebo/Bapineuzumab 0.5 mg/kg | Bapineuzumab 0.5 mg/kg/ Bapineuzumab 0.5 mg/kg | Placebo/Bapineuzumab 1.0 mg/kg | Bapineuzumab 1.0 mg/kg/Bapineuzumab 1.0 mg/kg | Bapineuzumab 2.0 mg/kg/ Bapineuzumab 1.0 mg/kg
Number analyzed (Participants) | 39 | 66 | 37 | 56 | 4
Number of participants | 6 | 10 | 1 | 11 | 0

2. Secondary Outcome: Change From Base Study Baseline in Alzheimer's Disease Assesment Scale-Cognitive Subscale (ADAS-Cog/11) at Weeks 13, 26, 39, 52 and 78.
Description: The ADAS-Cog is a multi-item, objective measure of cognitive function. The scale evaluates memory, language, and praxis with items such as orientation, word recall, word recognition, object identification, comprehension, and the completion of simple tasks. Analysis of the ADAS-Cog for this study was based upon an 11 item score from the following items 1) word recall task, 2) naming objects and fingers, 3) following commands, 4) constructional praxis, 5) ideational praxis, 6) orientation, 7) word recognition, 8) remembering test instructions, 9) spoken language ability, 10) word finding difficulty in spontaneous speech, and 11) comprehension.This scale had to be administered by a trained and certified psychometric rater who did not have access to any information regarding adverse events experienced. The ADAS-Cog/11 ranged from 0 to 70 points, with higher scores indicating a greater degree of impairment. A negative change from baseline indicates a decrease in cognitive impairment.
Time Frame: Weeks 13, 26, 39, 52 and 78
Population: The Extension mITT Population was defined as all randomly assigned participants who received at least one dose of investigational product in the extension study and who had a baseline for the extension study and at least one valid post-baseline assessment of the ADAS-Cog total score and DAD total score in the extension study.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo/Bapineuzumab 0.5 mg/kg | Bapineuzumab 0.5 mg/kg/ Bapineuzumab 0.5 mg/kg | Placebo/Bapineuzumab 1.0 mg/kg | Bapineuzumab 1.0 mg/kg/Bapineuzumab 1.0 mg/kg
Number analyzed (Participants) | 38 | 62 | 33 | 53
Units on a scale
  Week 13 (N = 38, 62, 33, 53) | 7.47 (1.17) | 6.17 (0.95) | 4.66 (1.26) | 6.45 (0.98)
  Week 26 (N = 33, 54, 26, 45) | 9.00 (1.27) | 7.49 (1.03) | 7.34 (1.38) | 7.30 (1.07)
  Week 39 (N = 25, 46, 22, 37) | 9.74 (1.35) | 8.79 (1.08) | 7.92 (1.45) | 9.50 (1.12)
  Week 52 (N = 18, 32, 15, 29) | 12.44 (1.70) | 10.38 (1.35) | 10.54 (1.82) | 10.31 (1.36)
  Week 78 (N = 12, 19, 8, 20) | 14.71 (2.12) | 12.27 (1.81) | 15.46 (2.46) | 15.31 (1.68)
Statistical Analysis 1: Comparison: Placebo/Bapineuzumab 0.5 mg/kg vs Bapineuzumab 0.5 mg/kg/ Bapineuzumab 0.5 mg/kg; Change from base study baseline in ADAS-Cog score at Week 13. Results are from a restricted maximum likelihood (REML)-based mixed model for repeated measures (MMRM) with change from base study baseline as the response and the following fixed effect model terms: treatment, visit (scheduled week), treatment-by-visit interaction, baseline value of the response variable, baseline MMSE total score stratum and cholinesterase inhibitor or memantine use stratum; Test type: Superiority or Other; p = 0.390, Mixed Models Analysis; Mean Difference (Final Values) = -1.30, 95% CI 2-sided [-4.29 to 1.68]
Statistical Analysis 2: Comparison: Placebo/Bapineuzumab 1.0 mg/kg vs Bapineuzumab 1.0 mg/kg/Bapineuzumab 1.0 mg/kg; Change from base study baseline in ADAS-Cog score at Week 13. Results are from a REML-based MMRM with change from base study baseline as the response and the following fixed effect model terms: treatment, visit (scheduled week), treatment-by-visit interaction, baseline value of the response variable, baseline MMSE total score stratum and cholinesterase inhibitor or memantine use stratum; Test type: Superiority or Other; p = 0.264, Mixed Models Analysis; Mean Difference (Final Values) = 1.80, 95% CI 2-sided [-1.37 to 4.97]
Statistical Analysis 3: Comparison: Placebo/Bapineuzumab 0.5 mg/kg vs Bapineuzumab 0.5 mg/kg/ Bapineuzumab 0.5 mg/kg; Change from base study baseline in ADAS-Cog score at Week 26. Results are from a REML-based MMRM with change from base study baseline as the response and the following fixed effect model terms: treatment, visit (scheduled week), treatment-by-visit interaction, baseline value of the response variable, baseline MMSE total score stratum and cholinesterase inhibitor or memantine use stratum; Test type: Superiority or Other; p = 0.357, Mixed Models Analysis; Mean Difference (Final Values) = -1.51, 95% CI 2-sided [-4.74 to 1.72]
Statistical Analysis 4: Comparison: Placebo/Bapineuzumab 1.0 mg/kg vs Bapineuzumab 1.0 mg/kg/Bapineuzumab 1.0 mg/kg; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.981, Mixed Models Analysis; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-3.50 to 3.42]
Statistical Analysis 5: Comparison: Placebo/Bapineuzumab 0.5 mg/kg vs Bapineuzumab 0.5 mg/kg/ Bapineuzumab 0.5 mg/kg; Change from base study baseline in ADAS-Cog score at Week 39. Results are from a REML-based MMRM with change from base study baseline as the response and the following fixed effect model terms: treatment, visit (scheduled week), treatment-by-visit interaction, baseline value of the response variable, baseline MMSE total score stratum and cholinesterase inhibitor or memantine use stratum; Test type: Superiority or Other; p = 0.584, Mixed Models Analysis; Mean Difference (Final Values) = -0.95, 95% CI 2-sided [-4.37 to 2.47]
Statistical Analysis 6: Comparison: Placebo/Bapineuzumab 1.0 mg/kg vs Bapineuzumab 1.0 mg/kg/Bapineuzumab 1.0 mg/kg; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.392, Mixed Models Analysis; Mean Difference (Final Values) = 1.58, 95% CI 2-sided [-2.05 to 5.20]
Statistical Analysis 7: Comparison: Placebo/Bapineuzumab 0.5 mg/kg vs Bapineuzumab 0.5 mg/kg/ Bapineuzumab 0.5 mg/kg; Change from base study baseline in ADAS-Cog score at Week 52. Results are from a REML-based MMRM with change from base study baseline as the response and the following fixed effect model terms: treatment, visit (scheduled week), treatment-by-visit interaction, baseline value of the response variable, baseline MMSE total score stratum and cholinesterase inhibitor or memantine use stratum; Test type: Superiority or Other; p = 0.345, Mixed Models Analysis; Mean Difference (Final Values) = -2.05, 95% CI 2-sided [-6.34 to 2.24]
Statistical Analysis 8: Comparison: Placebo/Bapineuzumab 1.0 mg/kg vs Bapineuzumab 1.0 mg/kg/Bapineuzumab 1.0 mg/kg; [analysis description as in outcome 2, analysis 7]; Test type: Superiority or Other; p = 0.922, Mixed Models Analysis; Mean Difference (Final Values) = -0.22, 95% CI 2-sided [-4.73 to 4.28]
Statistical Analysis 9: Comparison: Placebo/Bapineuzumab 0.5 mg/kg vs Bapineuzumab 0.5 mg/kg/ Bapineuzumab 0.5 mg/kg; Change from base study baseline in ADAS-Cog score at Week 78. Results are from a REML-based MMRM with change from base study baseline as the response and the following fixed effect model terms: treatment, visit (scheduled week), treatment-by-visit interaction, baseline value of the response variable, baseline MMSE total score stratum and cholinesterase inhibitor or memantine use stratum; Test type: Superiority or Other; p = 0.384, Mixed Models Analysis; Mean Difference (Final Values) = -2.44, 95% CI 2-sided [-7.97 to 3.10]
Statistical Analysis 10: Comparison: Placebo/Bapineuzumab 1.0 mg/kg vs Bapineuzumab 1.0 mg/kg/Bapineuzumab 1.0 mg/kg; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.961, Mixed Models Analysis; Mean Difference (Final Values) = -0.15, 95% CI 2-sided [-6.08 to 5.78]

3. Secondary Outcome: Change From Extension Study Baseline in ADAS-Cog/11 at Weeks 13, 26, 39, 52 and 78.
Description: as for outcome 2
Time Frame: Weeks 13, 26, 39, 52 and 78
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo/Bapineuzumab 0.5 mg/kg | Bapineuzumab 0.5 mg/kg/ Bapineuzumab 0.5 mg/kg | Placebo/Bapineuzumab 1.0 mg/kg | Bapineuzumab 1.0 mg/kg/Bapineuzumab 1.0 mg/kg
Number analyzed (Participants) | 38 | 62 | 33 | 53
Units on a scale
  Week 13 (N = 38, 62, 33, 53) | 0.10 (0.84) | 0.32 (0.68) | -1.68 (0.90) | 0.46 (0.70)
  Week 26 (N = 33, 54, 26, 45) | 1.61 (0.92) | 1.63 (0.75) | 1.08 (1.01) | 1.37 (0.78)
  Week 39 (N = 25, 46, 22, 37) | 2.35 (1.01) | 2.86 (0.79) | 1.68 (1.07) | 3.62 (0.83)
  Week 52 (N = 18, 32, 15, 29) | 4.85 (1.45) | 4.45 (1.14) | 4.30 (1.55) | 4.43 (1.14)
  Week 78 (N = 12, 19, 8, 20) | 7.29 (1.81) | 6.73 (1.57) | 8.86 (2.15) | 9.68 (1.42)
Statistical Analysis 1: Comparison: Placebo/Bapineuzumab 0.5 mg/kg vs Bapineuzumab 0.5 mg/kg/ Bapineuzumab 0.5 mg/kg; Change from extension study baseline in ADAS-Cog score at Week 13. Results are from a REML based MMRM with change from extension study baseline as the response and the following fixed effect model terms: treatment, visit (scheduled week), treatment-by-visit interaction, baseline value of the response variable, baseline MMSE total score stratum and cholinesterase inhibitor or memantine use stratum; Test type: Superiority or Other; p = 0.837, Mixed Models Analysis; Mean Difference (Final Values) = 0.22, 95% CI 2-sided [-1.91 to 2.35]
Statistical Analysis 2: Comparison: Placebo/Bapineuzumab 1.0 mg/kg vs Bapineuzumab 1.0 mg/kg/Bapineuzumab 1.0 mg/kg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.064, Mixed Models Analysis; Mean Difference (Final Values) = 2.14, 95% CI 2-sided [-0.13 to 4.41]
Statistical Analysis 3: Comparison: Placebo/Bapineuzumab 0.5 mg/kg vs Bapineuzumab 0.5 mg/kg/ Bapineuzumab 0.5 mg/kg; Change from extension study baseline in ADAS-Cog score at Week 26. Results are from a REML based MMRM with change from extension study baseline as the response and the following fixed effect model terms: treatment, visit (scheduled week), treatment-by-visit interaction, baseline value of the response variable, baseline MMSE total score stratum and cholinesterase inhibitor or memantine use stratum; Test type: Superiority or Other; p = 0.990, Mixed Models Analysis; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-2.32 to 2.35]
Statistical Analysis 4: Comparison: Placebo/Bapineuzumab 1.0 mg/kg vs Bapineuzumab 1.0 mg/kg/Bapineuzumab 1.0 mg/kg; [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; p = 0.817, Mixed Models Analysis; Mean Difference (Final Values) = 0.30, 95% CI 2-sided [-2.22 to 2.82]
Statistical Analysis 5: Comparison: Placebo/Bapineuzumab 0.5 mg/kg vs Bapineuzumab 0.5 mg/kg/ Bapineuzumab 0.5 mg/kg; Change from extension study baseline in ADAS-Cog score at Week 39. Results are from a REML based MMRM with change from extension study baseline as the response and the following fixed effect model terms: treatment, visit (scheduled week), treatment-by-visit interaction, baseline value of the response variable, baseline MMSE total score stratum and cholinesterase inhibitor or memantine use stratum; Test type: Superiority or Other; p = 0.697, Mixed Models Analysis; Mean Difference (Final Values) = 0.50, 95% CI 2-sided [-2.04 to 3.05]
Statistical Analysis 6: Comparison: Placebo/Bapineuzumab 1.0 mg/kg vs Bapineuzumab 1.0 mg/kg/Bapineuzumab 1.0 mg/kg; [analysis description as in outcome 3, analysis 5]; Test type: Superiority or Other; p = 0.158, Mixed Models Analysis; Mean Difference (Final Values) = 1.93, 95% CI 2-sided [-0.76 to 4.63]
Statistical Analysis 7: Comparison: Placebo/Bapineuzumab 0.5 mg/kg vs Bapineuzumab 0.5 mg/kg/ Bapineuzumab 0.5 mg/kg; Change from extension study baseline in ADAS-Cog score at Week 52. Results are from a REML based MMRM with change from extension study baseline as the response and the following fixed effect model terms: treatment, visit (scheduled week), treatment-by-visit interaction, baseline value of the response variable, baseline MMSE total score stratum and cholinesterase inhibitor or memantine use stratum; Test type: Superiority or Other; p = 0.829, Mixed Models Analysis; Mean Difference (Final Values) = -0.40, 95% CI 2-sided [-4.06 to 3.26]
Statistical Analysis 8: Comparison: Placebo/Bapineuzumab 1.0 mg/kg vs Bapineuzumab 1.0 mg/kg/Bapineuzumab 1.0 mg/kg; [analysis description as in outcome 3, analysis 7]; Test type: Superiority or Other; p = 0.950, Mixed Models Analysis; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [-3.69 to 3.93]
Statistical Analysis 9: Comparison: Placebo/Bapineuzumab 0.5 mg/kg vs Bapineuzumab 0.5 mg/kg/ Bapineuzumab 0.5 mg/kg; Change from extension study baseline in ADAS-Cog score at Week 78. Results are from a REML based MMRM with change from extension study baseline as the response and the following fixed effect model terms: treatment, visit (scheduled week), treatment-by-visit interaction, baseline value of the response variable, baseline MMSE total score stratum and cholinesterase inhibitor or memantine use stratum; Test type: Superiority or Other; p = 0.816, Mixed Models Analysis; Mean Difference (Final Values) = -0.56, 95% CI 2-sided [-5.35 to 4.23]
Statistical Analysis 10: Comparison: Placebo/Bapineuzumab 1.0 mg/kg vs Bapineuzumab 1.0 mg/kg/Bapineuzumab 1.0 mg/kg; [analysis description as in outcome 3, analysis 9]; Test type: Superiority or Other; p = 0.751, Mixed Models Analysis; Mean Difference (Final Values) = 0.82, 95% CI 2-sided [-4.32 to 5.96]

4. Secondary Outcome: Change From Base Study Baseline in Disability Assessment for Dementia (DAD) Score at Weeks 13, 26, 39, 52 and 78.
Description: The DAD measures instrumental and basic activities of daily living in participants with Alzheimer's Disease (AD). The DAD is administered to the participants'caregiver in the form of an interview. This scale had to be administered by a trained and certified psychometric rater who did not have access to any information regarding adverse events experienced by the participant. This scale assesses a participants' ability to initiate, plan, and perform activities related to hygiene, dressing, continence, eating, meal preparation, telephoning, going on an outing, finance and correspondence, medications, leisure, and housework. Each item can be scored as 1 = yes, 0 = no, non applicable = NA. A total score is obtained by adding the rating for each question and converting this total score out of 100. Higher scores indicate better function; a positive change from baseline indicates an improvement
Time Frame: Weeks 13, 26, 39, 52 and 78
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo/Bapineuzumab 0.5 mg/kg | Bapineuzumab 0.5 mg/kg/ Bapineuzumab 0.5 mg/kg | Placebo/Bapineuzumab 1.0 mg/kg | Bapineuzumab 1.0 mg/kg/Bapineuzumab 1.0 mg/kg
Number analyzed (Participants) | 38 | 62 | 33 | 53
Units on a scale
  Week 13 (N = 38, 62, 31, 52) | -18.75 (2.88) | -18.60 (2.36) | -15.50 (3.13) | -13.36 (2.43)
  Week 26 (N = 33, 56, 26, 44) | -21.19 (2.93) | -21.04 (2.38) | -16.26 (3.19) | -19.18 (2.48)
  Week 39 (N = 25, 46, 21, 37) | -25.42 (3.14) | -27.36 (2.51) | -14.57 (3.39) | -19.10 (2.62)
  Week 52 (N = 18, 32, 15, 30) | -29.52 (3.48) | -28.00 (2.77) | -20.41 (3.74) | -23.21 (2.80)
  Week 78 (N = 12, 20, 8, 20) | -36.48 (4.56) | -35.75 (3.79) | -25.21 (5.24) | -30.28 (3.65)
Statistical Analysis 1: Comparison: Placebo/Bapineuzumab 0.5 mg/kg vs Bapineuzumab 0.5 mg/kg/ Bapineuzumab 0.5 mg/kg; Change from base study baseline in DAD score at Week 13. Results are from a REML-based MMRM with change from base study baseline as the response and the following fixed effect model terms: treatment, visit (scheduled week), treatment-by-visit interaction, baseline value of the response variable, baseline MMSE total score stratum and cholinesterase inhibitor or memantine use stratum; Test type: Superiority or Other; p = 0.967, Mixed Models Analysis; Mean Difference (Final Values) = 0.16, 95% CI 2-sided [-7.22 to 7.53]
Statistical Analysis 2: Comparison: Placebo/Bapineuzumab 1.0 mg/kg vs Bapineuzumab 1.0 mg/kg/Bapineuzumab 1.0 mg/kg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.593, Mixed Models Analysis; Mean Difference (Final Values) = 2.13, 95% CI 2-sided [-5.72 to 9.98]
Statistical Analysis 3: Comparison: Placebo/Bapineuzumab 0.5 mg/kg vs Bapineuzumab 0.5 mg/kg/ Bapineuzumab 0.5 mg/kg; Change from base study baseline in DAD score at Week 26. Results are from a REML-based MMRM with change from base study baseline as the response and the following fixed effect model terms: treatment, visit (scheduled week), treatment-by-visit interaction, baseline value of the response variable, baseline MMSE total score stratum and cholinesterase inhibitor or memantine use stratum; Test type: Superiority or Other; p = 0.968, Mixed Models Analysis; Mean Difference (Final Values) = 0.15, 95% CI 2-sided [-7.32 to 7.62]
Statistical Analysis 4: Comparison: Placebo/Bapineuzumab 1.0 mg/kg vs Bapineuzumab 1.0 mg/kg/Bapineuzumab 1.0 mg/kg; [analysis description as in outcome 4, analysis 3]; Test type: Superiority or Other; p = 0.473, Mixed Models Analysis; Mean Difference (Final Values) = -2.92, 95% CI 2-sided [-10.92 to 5.08]
Statistical Analysis 5: Comparison: Placebo/Bapineuzumab 0.5 mg/kg vs Bapineuzumab 0.5 mg/kg/ Bapineuzumab 0.5 mg/kg; Change from base study baseline in DAD score at Week 39. Results are from a REML-based MMRM with change from base study baseline as the response and the following fixed effect model terms: treatment, visit (scheduled week), treatment-by-visit interaction, baseline value of the response variable, baseline MMSE total score stratum and cholinesterase inhibitor or memantine use stratum; Test type: Superiority or Other; p = 0.630, Mixed Models Analysis; Mean Difference (Final Values) = -1.95, 95% CI 2-sided [-9.91 to 6.02]
Statistical Analysis 6: Comparison: Placebo/Bapineuzumab 1.0 mg/kg vs Bapineuzumab 1.0 mg/kg/Bapineuzumab 1.0 mg/kg; [analysis description as in outcome 4, analysis 5]; Test type: Superiority or Other; p = 0.293, Mixed Models Analysis; Mean Difference (Final Values) = -4.53, 95% CI 2-sided [-13.02 to 3.95]
Statistical Analysis 7: Comparison: Placebo/Bapineuzumab 0.5 mg/kg vs Bapineuzumab 0.5 mg/kg/ Bapineuzumab 0.5 mg/kg; Change from base study baseline in DAD score at Week 52. Results are from a REML-based MMRM with change from base study baseline as the response and the following fixed effect model terms: treatment, visit (scheduled week), treatment-by-visit interaction, baseline value of the response variable, baseline MMSE total score stratum and cholinesterase inhibitor or memantine use stratum; Test type: Superiority or Other; p = 0.733, Mixed Models Analysis; Mean Difference (Final Values) = 1.53, 95% CI 2-sided [-7.28 to 10.33]
Statistical Analysis 8: Comparison: Placebo/Bapineuzumab 1.0 mg/kg vs Bapineuzumab 1.0 mg/kg/Bapineuzumab 1.0 mg/kg; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p = 0.550, Mixed Models Analysis; Mean Difference (Final Values) = -2.81, 95% CI 2-sided [-12.06 to 6.45]
Statistical Analysis 9: Comparison: Placebo/Bapineuzumab 0.5 mg/kg vs Bapineuzumab 0.5 mg/kg/ Bapineuzumab 0.5 mg/kg; Change from base study baseline in DAD score at Week 78. Results are from a REML-based MMRM with change from base study baseline as the response and the following fixed effect model terms: treatment, visit (scheduled week), treatment-by-visit interaction, baseline value of the response variable, baseline MMSE total score stratum and cholinesterase inhibitor or memantine use stratum; Test type: Superiority or Other; p = 0.902, Mixed Models Analysis; Mean Difference (Final Values) = 0.73, 95% CI 2-sided [-11.04 to 12.50]
Statistical Analysis 10: Comparison: Placebo/Bapineuzumab 1.0 mg/kg vs Bapineuzumab 1.0 mg/kg/Bapineuzumab 1.0 mg/kg; [analysis description as in outcome 4, analysis 9]; Test type: Superiority or Other; p = 0.430, Mixed Models Analysis; Mean Difference (Final Values) = -5.07, 95% CI 2-sided [-17.75 to 7.61]

5. Secondary Outcome: Change From Extension Study Baseline in DAD Score at Weeks 13, 26, 39, 52 and 78
Description: The DAD measures instrumental and basic activities of daily living in participants with AD. The DAD is administered to the participants'caregiver in the form of an interview. This scale had to be administered by a trained and certified psychometric rater who did not have access to any information regarding adverse events experienced by the participant. This scale assesses a participants' ability to initiate, plan, and perform activities related to hygiene, dressing, continence, eating, meal preparation, telephoning, going on an outing, finance and correspondence, medications, leisure, and housework. Each item can be scored as 1 = yes, 0 = no, non applicable = NA. A total score is obtained by adding the rating for each question and converting this total score out of 100. Higher scores indicate better function; a positive change from baseline indicates an improvement
Time Frame: Weeks 13, 26, 39, 52 and 78
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo/Bapineuzumab 0.5 mg/kg | Bapineuzumab 0.5 mg/kg/ Bapineuzumab 0.5 mg/kg | Placebo/Bapineuzumab 1.0 mg/kg | Bapineuzumab 1.0 mg/kg/Bapineuzumab 1.0 mg/kg
Number analyzed (Participants) | 38 | 62 | 33 | 53
Units on a scale
  Week 13 (N = 38, 62, 31, 52) | -3.80 (1.96) | -4.83 (1.60) | -5.17 (2.16) | -1.48 (1.65)
  Week 26 (N = 33, 56, 26, 44) | -6.33 (2.02) | -7.22 (1.64) | -5.75 (2.23) | -7.25 (1.73)
  Week 39 (N = 25, 46, 21, 37) | -11.14 (2.23) | -13.49 (1.76) | -4.34 (2.41) | -7.08 (1.85)
  Week 52 (N = 18, 32, 15, 30) | -16.21 (2.57) | -13.77 (2.02) | -10.02 (2.75) | -11.06 (2.02)
  Week 78 (N = 12, 20, 8, 20) | -23.40 (3.01) | -21.30 (2.54) | -14.54 (3.54) | -17.41 (2.37)
Statistical Analysis 1: Comparison: Placebo/Bapineuzumab 0.5 mg/kg vs Bapineuzumab 0.5 mg/kg/ Bapineuzumab 0.5 mg/kg; Change from extension study baseline in DAD score at Week 13. Results are from a REML based MMRM with change from extension study baseline as the response and the following fixed effect model terms: treatment, visit (scheduled week), treatment-by-visit interaction, baseline value of the response variable, baseline MMSE total score stratum and cholinesterase inhibitor or memantine use stratum; Test type: Superiority or Other; p = 0.683, Mixed Models Analysis; Mean Difference (Final Values) = -1.03, 95% CI 2-sided [-6.01 to 3.95]
Statistical Analysis 2: Comparison: Placebo/Bapineuzumab 1.0 mg/kg vs Bapineuzumab 1.0 mg/kg/Bapineuzumab 1.0 mg/kg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.177, Mixed Models Analysis; Mean Difference (Final Values) = 3.69, 95% CI 2-sided [-1.68 to 9.06]
Statistical Analysis 3: Comparison: Placebo/Bapineuzumab 0.5 mg/kg vs Bapineuzumab 0.5 mg/kg/ Bapineuzumab 0.5 mg/kg; Change from extension study baseline in DAD score at Week 26. Results are from a REML based MMRM with change from extension study baseline as the response and the following fixed effect model terms: treatment, visit (scheduled week), treatment-by-visit interaction, baseline value of the response variable, baseline MMSE total score stratum and cholinesterase inhibitor or memantine use stratum; Test type: Superiority or Other; p = 0.734, Mixed Models Analysis; Mean Difference (Final Values) = -0.89, 95% CI 2-sided [-6.03 to 4.25]
Statistical Analysis 4: Comparison: Placebo/Bapineuzumab 1.0 mg/kg vs Bapineuzumab 1.0 mg/kg/Bapineuzumab 1.0 mg/kg; [analysis description as in outcome 5, analysis 3]; Test type: Superiority or Other; p = 0.595, Mixed Models Analysis; Mean Difference (Final Values) = -1.50, 95% CI 2-sided [-7.06 to 4.05]
Statistical Analysis 5: Comparison: Placebo/Bapineuzumab 0.5 mg/kg vs Bapineuzumab 0.5 mg/kg/ Bapineuzumab 0.5 mg/kg; Change from extension study baseline in DAD score at Week 39. Results are from a REML based MMRM with change from extension study baseline as the response and the following fixed effect model terms: treatment, visit (scheduled week), treatment-by-visit interaction, baseline value of the response variable, baseline MMSE total score stratum and cholinesterase inhibitor or memantine use stratum; Test type: Superiority or Other; p = 0.409, Mixed Models Analysis; Mean Difference (Final Values) = -2.35, 95% CI 2-sided [-7.95 to 3.24]
Statistical Analysis 6: Comparison: Placebo/Bapineuzumab 1.0 mg/kg vs Bapineuzumab 1.0 mg/kg/Bapineuzumab 1.0 mg/kg; [analysis description as in outcome 5, analysis 5]; Test type: Superiority or Other; p = 0.368, Mixed Models Analysis; Mean Difference (Final Values) = -2.74, 95% CI 2-sided [-8.73 to 3.24]
Statistical Analysis 7: Comparison: Placebo/Bapineuzumab 0.5 mg/kg vs Bapineuzumab 0.5 mg/kg/ Bapineuzumab 0.5 mg/kg; Change from extension study baseline in DAD score at Week 52. Results are from a REML based MMRM with change from extension study baseline as the response and the following fixed effect model terms: treatment, visit (scheduled week), treatment-by-visit interaction, baseline value of the response variable, baseline MMSE total score stratum and cholinesterase inhibitor or memantine use stratum; Test type: Superiority or Other; p = 0.458, Mixed Models Analysis; Mean Difference (Final Values) = 2.44, 95% CI 2-sided [-4.01 to 8.89]
Statistical Analysis 8: Comparison: Placebo/Bapineuzumab 1.0 mg/kg vs Bapineuzumab 1.0 mg/kg/Bapineuzumab 1.0 mg/kg; [analysis description as in outcome 5, analysis 7]; Test type: Superiority or Other; p = 0.760, Mixed Models Analysis; Mean Difference (Final Values) = -1.04, 95% CI 2-sided [-7.77 to 5.68]
Statistical Analysis 9: Comparison: Placebo/Bapineuzumab 0.5 mg/kg vs Bapineuzumab 0.5 mg/kg/ Bapineuzumab 0.5 mg/kg; Change from extension study baseline in DAD score at Week 78. Results are from a REML based MMRM with change from extension study baseline as the response and the following fixed effect model terms: treatment, visit (scheduled week), treatment-by-visit interaction, baseline value of the response variable, baseline MMSE total score stratum and cholinesterase inhibitor or memantine use stratum; Test type: Superiority or Other; p = 0.597, Mixed Models Analysis; Mean Difference (Final Values) = 2.09, 95% CI 2-sided [-5.67 to 9.86]
Statistical Analysis 10: Comparison: Placebo/Bapineuzumab 1.0 mg/kg vs Bapineuzumab 1.0 mg/kg/Bapineuzumab 1.0 mg/kg; [analysis description as in outcome 5, analysis 9]; Test type: Superiority or Other; p = 0.501, Mixed Models Analysis; Mean Difference (Final Values) = -2.87, 95% CI 2-sided [-11.24 to 5.50]

6. Secondary Outcome: Change From Base Study Baseline in Neuropsychiatric Inventory (NPI) Score at Weeks 26, 52 and 78.
Description: NPI:12-domain caregiver assessment of behavioral disturbances occurring in dementia: delusions, hallucinations, agitation/aggression, depression/dysphoria, anxiety, elation/euphoria, apathy/indifference, disinhibition, irritability/lability, motor disturbance, appetite/eating, nighttime behavior. Severity (1=Mild to 3=Severe), frequency (1=occasionally to 4=very frequently) scales recorded for each domain; frequency*severity=each domain score(range 0-12). Total score=sum of each domain score (range 0-144); higher score=greater behavioral disturbances; negative change score from baseline=improvement.
Time Frame: Weeks 26, 52 and 78
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo/Bapineuzumab 0.5 mg/kg | Bapineuzumab 0.5 mg/kg/ Bapineuzumab 0.5 mg/kg | Placebo/Bapineuzumab 1.0 mg/kg | Bapineuzumab 1.0 mg/kg/Bapineuzumab 1.0 mg/kg
Number analyzed (Participants) | 38 | 62 | 33 | 53
Units on a scale
  Week 26 (N = 36, 59, 30, 51) | 4.57 (2.08) | 0.97 (1.70) | 4.71 (2.26) | 4.43 (1.75)
  Week 52 (N = 21, 37, 17, 32) | 4.99 (2.60) | -0.01 (2.05) | 4.23 (2.80) | 6.57 (2.08)
  Week 78 (N = 13, 18, 8, 20) | 16.17 (3.23) | 3.31 (2.94) | 5.24 (4.02) | 6.70 (2.61)
Statistical Analysis 1: Comparison: Placebo/Bapineuzumab 0.5 mg/kg vs Bapineuzumab 0.5 mg/kg/ Bapineuzumab 0.5 mg/kg; Change from base study baseline in NPI score at Week 26. Results are from a REML-based MMRM with change from base study baseline as the response and the following fixed effect model terms: treatment, visit (scheduled week), treatment-by-visit interaction, baseline value of the response variable, baseline MMSE total score stratum and cholinesterase inhibitor or memantine use stratum; Test type: Superiority or Other; p = 0.183, Mixed Models Analysis; Mean Difference (Final Values) = -3.60, 95% CI 2-sided [-8.91 to 1.71]
Statistical Analysis 2: Comparison: Placebo/Bapineuzumab 1.0 mg/kg vs Bapineuzumab 1.0 mg/kg/Bapineuzumab 1.0 mg/kg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.920, Mixed Models Analysis; Mean Difference (Final Values) = -0.29, 95% CI 2-sided [-5.92 to 5.35]
Statistical Analysis 3: Comparison: Placebo/Bapineuzumab 0.5 mg/kg vs Bapineuzumab 0.5 mg/kg/ Bapineuzumab 0.5 mg/kg; Change from base study baseline in NPI score at Week 52. Results are from a REML-based MMRM with change from base study baseline as the response and the following fixed effect model terms: treatment, visit (scheduled week), treatment-by-visit interaction, baseline value of the response variable, baseline MMSE total score stratum and cholinesterase inhibitor or memantine use stratum; Test type: Superiority or Other; p = 0.133, Mixed Models Analysis; Mean Difference (Final Values) = -4.99, 95% CI 2-sided [-11.52 to 1.53]
Statistical Analysis 4: Comparison: Placebo/Bapineuzumab 1.0 mg/kg vs Bapineuzumab 1.0 mg/kg/Bapineuzumab 1.0 mg/kg; [analysis description as in outcome 6, analysis 3]; Test type: Superiority or Other; p = 0.505, Mixed Models Analysis; Mean Difference (Final Values) = 2.34, 95% CI 2-sided [-4.55 to 9.22]
Statistical Analysis 5: Comparison: Placebo/Bapineuzumab 0.5 mg/kg vs Bapineuzumab 0.5 mg/kg/ Bapineuzumab 0.5 mg/kg; Change from base study baseline in NPI score at Week 78. Results are from a REML-based MMRM with change from base study baseline as the response and the following fixed effect model terms: treatment, visit (scheduled week), treatment-by-visit interaction, baseline value of the response variable, baseline MMSE total score stratum and cholinesterase inhibitor or memantine use stratum; Test type: Superiority or Other; p = 0.003, Mixed Models Analysis; Mean Difference (Final Values) = -12.86, 95% CI 2-sided [-21.46 to -4.25]
Statistical Analysis 6: Comparison: Placebo/Bapineuzumab 1.0 mg/kg vs Bapineuzumab 1.0 mg/kg/Bapineuzumab 1.0 mg/kg; [analysis description as in outcome 6, analysis 5]; Test type: Superiority or Other; p = 0.760, Mixed Models Analysis; Mean Difference (Final Values) = 1.47, 95% CI 2-sided [-7.95 to 10.88]

7. Secondary Outcome: Change From Extension Study Baseline in NPI Score at Weeks 26, 52 and 78.
Description: NPI:12-domain caregiver assessment of behavioral disturbances occurring in dementia: delusions, hallucinations, agitation/aggression, depression/dysphoria, anxiety, elation/euphoria, apathy/indifference, disinhibition, irritability/lability, motor disturbance, appetite/eating, night-time behavior. Severity (1=Mild to 3=Severe), frequency (1=occasionally to 4=very frequently) scales recorded for each domain; frequency*severity=each domain score(range 0-12). Total score=sum of each domain score(range 0-144); higher score=greater behavioral disturbances; negative change score from baseline=improvement.
Time Frame: Weeks 26, 52 and 78
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo/Bapineuzumab 0.5 mg/kg | Bapineuzumab 0.5 mg/kg/ Bapineuzumab 0.5 mg/kg | Placebo/Bapineuzumab 1.0 mg/kg | Bapineuzumab 1.0 mg/kg/Bapineuzumab 1.0 mg/kg
Number analyzed (Participants) | 38 | 62 | 33 | 53
Units on a scale
  Week 26 (N = 36, 60, 30, 51) | 2.29 (1.79) | 0.21 (1.48) | 2.77 (1.96) | 1.73 (1.51)
  Week 52 (N = 21, 37, 17, 32) | 2.34 (2.45) | -1.06 (1.94) | 3.78 (2.65) | 3.99 (1.97)
  Week 78 (N = 13, 18, 8, 20) | 11.76 (4.86) | 1.70 (4.40) | 2.28 (6.07) | 4.76 (3.93)
Statistical Analysis 1: Comparison: Placebo/Bapineuzumab 0.5 mg/kg vs Bapineuzumab 0.5 mg/kg/ Bapineuzumab 0.5 mg/kg; Change from extension study baseline in NPI score at Week 26. Results are from a REML based MMRM with change from extension study baseline as the response and the following fixed effect model terms: treatment, visit (scheduled week), treatment-by-visit interaction, baseline value of the response variable, baseline MMSE total score stratum and cholinesterase inhibitor or memantine use stratum; Test type: Superiority or Other; p = 0.373, Mixed Models Analysis; Mean Difference (Final Values) = -2.08, 95% CI 2-sided [-6.68 to 2.52]
Statistical Analysis 2: Comparison: Placebo/Bapineuzumab 1.0 mg/kg vs Bapineuzumab 1.0 mg/kg/Bapineuzumab 1.0 mg/kg; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.677, Mixed Models Analysis; Mean Difference (Final Values) = -1.03, 95% CI 2-sided [-5.92 to 3.86]
Statistical Analysis 3: Comparison: Placebo/Bapineuzumab 0.5 mg/kg vs Bapineuzumab 0.5 mg/kg/ Bapineuzumab 0.5 mg/kg; Change from extension study baseline in NPI score at Week 52. Results are from a REML based MMRM with change from extension study baseline as the response and the following fixed effect model terms: treatment, visit (scheduled week), treatment-by-visit interaction, baseline value of the response variable, baseline MMSE total score stratum and cholinesterase inhibitor or memantine use stratum; Test type: Superiority or Other; p = 0.280, Mixed Models Analysis; Mean Difference (Final Values) = -3.40, 95% CI 2-sided [-9.61 to 2.80]
Statistical Analysis 4: Comparison: Placebo/Bapineuzumab 1.0 mg/kg vs Bapineuzumab 1.0 mg/kg/Bapineuzumab 1.0 mg/kg; [analysis description as in outcome 7, analysis 3]; Test type: Superiority or Other; p = 0.950, Mixed Models Analysis; Mean Difference (Final Values) = 0.21, 95% CI 2-sided [-6.34 to 6.76]
Statistical Analysis 5: Comparison: Placebo/Bapineuzumab 0.5 mg/kg vs Bapineuzumab 0.5 mg/kg/ Bapineuzumab 0.5 mg/kg; Change from extension study baseline in NPI score at Week 78. Results are from a REML based MMRM with change from extension study baseline as the response and the following fixed effect model terms: treatment, visit (scheduled week), treatment-by-visit interaction, baseline value of the response variable, baseline MMSE total score stratum and cholinesterase inhibitor or memantine use stratum; Test type: Superiority or Other; p = 0.130, Mixed Models Analysis; Mean Difference (Final Values) = -10.06, 95% CI 2-sided [-23.16 to 3.05]
Statistical Analysis 6: Comparison: Placebo/Bapineuzumab 1.0 mg/kg vs Bapineuzumab 1.0 mg/kg/Bapineuzumab 1.0 mg/kg; [analysis description as in outcome 7, analysis 5]; Test type: Superiority or Other; p = 0.732, Mixed Models Analysis; Mean Difference (Final Values) = 2.48, 95% CI 2-sided [-11.97 to 16.94]

8. Secondary Outcome: Change From Base Study Baseline in Mini-mental State Examination (MMSE) Score at Weeks 6, 19, 32, 45 and 78.
Description: MMSE measured general cognitive functioning: orientation, memory, attention, concentration, naming, repetition, comprehension, and ability to create a sentence and to copy two intersecting polygons. Total score derived from sub-scores; total ranged from 0 to 30, higher score indicates better cognitive state.
Time Frame: Weeks 6, 19, 32, 45 and 78
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo/Bapineuzumab 0.5 mg/kg | Bapineuzumab 0.5 mg/kg/ Bapineuzumab 0.5 mg/kg | Placebo/Bapineuzumab 1.0 mg/kg | Bapineuzumab 1.0 mg/kg/Bapineuzumab 1.0 mg/kg
Number analyzed (Participants) | 38 | 62 | 33 | 53
Units on a scale
  Week 6 (N = 38, 61, 33, 53) | -2.89 (0.46) | -2.85 (0.37) | -2.02 (0.49) | -2.22 (0.39)
  Week 19 (N = 36, 59, 28, 50) | -2.80 (0.47) | -2.66 (0.38) | -2.76 (0.51) | -3.29 (0.39)
  Week 32 (N = 32, 51, 26, 41) | -3.82 (0.49) | -3.43 (0.40) | -4.40 (0.53) | -3.88 (0.42)
  Week 45 (N = 23, 41, 21, 35) | -4.86 (0.56) | -4.13 (0.44) | -4.63 (0.58) | -4.51 (0.46)
  Week 78 (N = 13, 27, 11, 21) | -7.62 (0.70) | -5.10 (0.54) | -6.97 (0.75) | -4.89 (0.56)
Statistical Analysis 1: Comparison: Placebo/Bapineuzumab 0.5 mg/kg vs Bapineuzumab 0.5 mg/kg/ Bapineuzumab 0.5 mg/kg; Change from base study baseline in MMSE score at Week 6. Results are from a REML-based MMRM with change from base study baseline as the response and the following fixed effect model terms: treatment, visit (scheduled week), treatment-by-visit interaction, baseline value of the response variable, baseline MMSE total score stratum and cholinesterase inhibitor or memantine use stratum; Test type: Superiority or Other; p = 0.938, Mixed Models Analysis; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [-1.12 to 1.21]
Statistical Analysis 2: Comparison: Placebo/Bapineuzumab 1.0 mg/kg vs Bapineuzumab 1.0 mg/kg/Bapineuzumab 1.0 mg/kg; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.753, Mixed Models Analysis; Mean Difference (Final Values) = -0.20, 95% CI 2-sided [-1.43 to 1.04]
Statistical Analysis 3: Comparison: Placebo/Bapineuzumab 0.5 mg/kg vs Bapineuzumab 0.5 mg/kg/ Bapineuzumab 0.5 mg/kg; Change from base study baseline in MMSE score at Week 19. Results are from a REML-based MMRM with change from base study baseline as the response and the following fixed effect model terms: treatment, visit (scheduled week), treatment-by-visit interaction, baseline value of the response variable, baseline MMSE total score stratum and cholinesterase inhibitor or memantine use stratum; Test type: Superiority or Other; p = 0.809, Mixed Models Analysis; Mean Difference (Final Values) = 0.15, 95% CI 2-sided [-1.04 to 1.33]
Statistical Analysis 4: Comparison: Placebo/Bapineuzumab 1.0 mg/kg vs Bapineuzumab 1.0 mg/kg/Bapineuzumab 1.0 mg/kg; [analysis description as in outcome 8, analysis 3]; Test type: Superiority or Other; p = 0.421, Mixed Models Analysis; Mean Difference (Final Values) = -0.52, 95% CI 2-sided [-1.80 to 0.75]
Statistical Analysis 5: Comparison: Placebo/Bapineuzumab 0.5 mg/kg vs Bapineuzumab 0.5 mg/kg/ Bapineuzumab 0.5 mg/kg; Change from base study baseline in MMSE score at Week 32. Results are from a REML-based MMRM with change from base study baseline as the response and the following fixed effect model terms: treatment, visit (scheduled week), treatment-by-visit interaction, baseline value of the response variable, baseline MMSE total score stratum and cholinesterase inhibitor or memantine use stratum; Test type: Superiority or Other; p = 0.535, Mixed Models Analysis; Mean Difference (Final Values) = 0.39, 95% CI 2-sided [-0.85 to 1.63]
Statistical Analysis 6: Comparison: Placebo/Bapineuzumab 1.0 mg/kg vs Bapineuzumab 1.0 mg/kg/Bapineuzumab 1.0 mg/kg; [analysis description as in outcome 8, analysis 5]; Test type: Superiority or Other; p = 0.445, Mixed Models Analysis; Mean Difference (Final Values) = 0.52, 95% CI 2-sided [-0.82 to 1.86]
Statistical Analysis 7: Comparison: Placebo/Bapineuzumab 0.5 mg/kg vs Bapineuzumab 0.5 mg/kg/ Bapineuzumab 0.5 mg/kg; Change from base study baseline in MMSE score at Week 45. Results are from a REML-based MMRM with change from base study baseline as the response and the following fixed effect model terms: treatment, visit (scheduled week), treatment-by-visit interaction, baseline value of the response variable, baseline MMSE total score stratum and cholinesterase inhibitor or memantine use stratum; Test type: Superiority or Other; p = 0.309, Mixed Models Analysis; Mean Difference (Final Values) = 0.73, 95% CI 2-sided [-0.67 to 2.12]
Statistical Analysis 8: Comparison: Placebo/Bapineuzumab 1.0 mg/kg vs Bapineuzumab 1.0 mg/kg/Bapineuzumab 1.0 mg/kg; [analysis description as in outcome 8, analysis 7]; Test type: Superiority or Other; p = 0.872, Mixed Models Analysis; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [-1.34 to 1.57]
Statistical Analysis 9: Comparison: Placebo/Bapineuzumab 0.5 mg/kg vs Bapineuzumab 0.5 mg/kg/ Bapineuzumab 0.5 mg/kg; Change from base study baseline in MMSE score at Week 78. Results are from a REML-based MMRM with change from base study baseline as the response and the following fixed effect model terms: treatment, visit (scheduled week), treatment-by-visit interaction, baseline value of the response variable, baseline MMSE total score stratum and cholinesterase inhibitor or memantine use stratum; Test type: Superiority or Other; p = 0.004, Mixed Models Analysis; Mean Difference (Final Values) = 2.52, 95% CI 2-sided [0.79 to 4.26]
Statistical Analysis 10: Comparison: Placebo/Bapineuzumab 1.0 mg/kg vs Bapineuzumab 1.0 mg/kg/Bapineuzumab 1.0 mg/kg; [analysis description as in outcome 8, analysis 9]; Test type: Superiority or Other; p = 0.026, Mixed Models Analysis; Mean Difference (Final Values) = 2.09, 95% CI 2-sided [0.25 to 3.93]

9. Secondary Outcome: Change From Extension Study Baseline in MMSE Score at Weeks 6, 19, 32, 45 and 78.
Description: as for outcome 8
Time Frame: Weeks 6, 19, 32, 45 and 78
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo/Bapineuzumab 0.5 mg/kg | Bapineuzumab 0.5 mg/kg/ Bapineuzumab 0.5 mg/kg | Placebo/Bapineuzumab 1.0 mg/kg | Bapineuzumab 1.0 mg/kg/Bapineuzumab 1.0 mg/kg
Number analyzed (Participants) | 38 | 62 | 33 | 53
Units on a scale
  Week 6 (N = 38, 61, 33, 53) | -1.20 (0.46) | -0.80 (0.38) | 0.11 (0.50) | -0.23 (0.39)
  Week 19 (N = 36, 59, 28, 50) | -1.10 (0.47) | -0.64 (0.38) | -0.62 (0.52) | -1.32 (0.39)
  Week 32 (N = 32, 51, 26, 41) | -2.11 (0.49) | -1.45 (0.40) | -2.18 (0.54) | -1.93 (0.42)
  Week 45 (N = 23, 41, 21, 35) | -3.06 (0.56) | -2.13 (0.45) | -2.39 (0.59) | -2.62 (0.46)
  Week 78 (N = 13, 27, 11, 21) | -5.68 (0.71) | -3.22 (0.54) | -4.73 (0.77) | -2.97 (0.56)
Statistical Analysis 1: Comparison: Placebo/Bapineuzumab 0.5 mg/kg vs Bapineuzumab 0.5 mg/kg/ Bapineuzumab 0.5 mg/kg; Change from extension study baseline in MMSE score at Week 6. Results are from a REML based MMRM with change from extension study baseline as the response and the following fixed effect model terms: treatment, visit (scheduled week), treatment-by-visit interaction, baseline value of the response variable, baseline MMSE total score stratum and cholinesterase inhibitor or memantine use stratum; Test type: Superiority or Other; p = 0.504, Mixed Models Analysis; Mean Difference (Final Values) = 0.40, 95% CI 2-sided [-0.77 to 1.57]
Statistical Analysis 2: Comparison: Placebo/Bapineuzumab 1.0 mg/kg vs Bapineuzumab 1.0 mg/kg/Bapineuzumab 1.0 mg/kg; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.592, Mixed Models Analysis; Mean Difference (Final Values) = -0.34, 95% CI 2-sided [-1.58 to 0.90]
Statistical Analysis 3: Comparison: Placebo/Bapineuzumab 0.5 mg/kg vs Bapineuzumab 0.5 mg/kg/ Bapineuzumab 0.5 mg/kg; Change from extension study baseline in MMSE score at Week 19. Results are from a REML based MMRM with change from extension study baseline as the response and the following fixed effect model terms: treatment, visit (scheduled week), treatment-by-visit interaction, baseline value of the response variable, baseline MMSE total score stratum and cholinesterase inhibitor or memantine use stratum; Test type: Superiority or Other; p = 0.441, Mixed Models Analysis; Mean Difference (Final Values) = 0.47, 95% CI 2-sided [-0.72 to 1.65]
Statistical Analysis 4: Comparison: Placebo/Bapineuzumab 1.0 mg/kg vs Bapineuzumab 1.0 mg/kg/Bapineuzumab 1.0 mg/kg; [analysis description as in outcome 9, analysis 3]; Test type: Superiority or Other; p = 0.288, Mixed Models Analysis; Mean Difference (Final Values) = -0.69, 95% CI 2-sided [-1.97 to 0.59]
Statistical Analysis 5: Comparison: Placebo/Bapineuzumab 0.5 mg/kg vs Bapineuzumab 0.5 mg/kg/ Bapineuzumab 0.5 mg/kg; Change from extension study baseline in MMSE score at Week 32. Results are from a REML based MMRM with change from extension study baseline as the response and the following fixed effect model terms: treatment, visit (scheduled week), treatment-by-visit interaction, baseline value of the response variable, baseline MMSE total score stratum and cholinesterase inhibitor or memantine use stratum; Test type: Superiority or Other; p = 0.303, Mixed Models Analysis; Mean Difference (Final Values) = 0.66, 95% CI 2-sided [-0.59 to 1.90]
Statistical Analysis 6: Comparison: Placebo/Bapineuzumab 1.0 mg/kg vs Bapineuzumab 1.0 mg/kg/Bapineuzumab 1.0 mg/kg; [analysis description as in outcome 9, analysis 5]; Test type: Superiority or Other; p = 0.713, Mixed Models Analysis; Mean Difference (Final Values) = 0.25, 95% CI 2-sided [-1.09 to 1.60]
Statistical Analysis 7: Comparison: Placebo/Bapineuzumab 0.5 mg/kg vs Bapineuzumab 0.5 mg/kg/ Bapineuzumab 0.5 mg/kg; Change from extension study baseline in MMSE score at Week 45. Results are from a REML based MMRM with change from extension study baseline as the response and the following fixed effect model terms: treatment, visit (scheduled week), treatment-by-visit interaction, baseline value of the response variable, baseline MMSE total score stratum and cholinesterase inhibitor or memantine use stratum; Test type: Superiority or Other; p = 0.198, Mixed Models Analysis; Mean Difference (Final Values) = 0.93, 95% CI 2-sided [-0.49 to 2.34]
Statistical Analysis 8: Comparison: Placebo/Bapineuzumab 1.0 mg/kg vs Bapineuzumab 1.0 mg/kg/Bapineuzumab 1.0 mg/kg; [analysis description as in outcome 9, analysis 7]; Test type: Superiority or Other; p = 0.756, Mixed Models Analysis; Mean Difference (Final Values) = -0.23, 95% CI 2-sided [-1.70 to 1.24]
Statistical Analysis 9: Comparison: Placebo/Bapineuzumab 0.5 mg/kg vs Bapineuzumab 0.5 mg/kg/ Bapineuzumab 0.5 mg/kg; Change from extension study baseline in MMSE score at Week 78. Results are from a REML based MMRM with change from extension study baseline as the response and the following fixed effect model terms: treatment, visit (scheduled week), treatment-by-visit interaction, baseline value of the response variable, baseline MMSE total score stratum and cholinesterase inhibitor or memantine use stratum; Test type: Superiority or Other; p = 0.006, Mixed Models Analysis; Mean Difference (Final Values) = 2.45, 95% CI 2-sided [0.69 to 4.22]
Statistical Analysis 10: Comparison: Placebo/Bapineuzumab 1.0 mg/kg vs Bapineuzumab 1.0 mg/kg/Bapineuzumab 1.0 mg/kg; [analysis description as in outcome 9, analysis 9]; Test type: Superiority or Other; p = 0.066, Mixed Models Analysis; Mean Difference (Final Values) = 1.75, 95% CI 2-sided [-0.12 to 3.62]

ADVERSE EVENTS:
Time Frame: 2.6 years
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Placebo/Bapineuzumab 0.5 mg/kg | Bapineuzumab 0.5 mg/kg/ Bapineuzumab 0.5 mg/kg | Placebo/Bapineuzumab 1.0 mg/kg | Bapineuzumab 1.0 mg/kg/Bapineuzumab 1.0 mg/kg | Bapineuzumab 2.0 mg/kg/Bapineuzumab 1.0 mg/kg
Serious Adverse Events (participants affected / at risk) | 6/39 | 10/66 | 1/37 | 11/56 | 0/4
Other Adverse Events (participants affected / at risk) | 18/39 | 21/66 | 15/37 | 15/56 | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo/Bapineuzumab 0.5 mg/kg (N=39) | Bapineuzumab 0.5 mg/kg/ Bapineuzumab 0.5 mg/kg (N=66) | Placebo/Bapineuzumab 1.0 mg/kg (N=37) | Bapineuzumab 1.0 mg/kg/Bapineuzumab 1.0 mg/kg (N=56) | Bapineuzumab 2.0 mg/kg/Bapineuzumab 1.0 mg/kg (N=4)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Chest injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebellar infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dementia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Partial seizures with secondary generalisation (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vasogenic cerebral oedema (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Disorientation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo/Bapineuzumab 0.5 mg/kg (N=39) | Bapineuzumab 0.5 mg/kg/ Bapineuzumab 0.5 mg/kg (N=66) | Placebo/Bapineuzumab 1.0 mg/kg (N=37) | Bapineuzumab 1.0 mg/kg/Bapineuzumab 1.0 mg/kg (N=56) | Bapineuzumab 2.0 mg/kg/Bapineuzumab 1.0 mg/kg (N=4)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arteriosclerotic retinopathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (3) | 1 (1) | 1 (2) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 7 (7) | 1 (2) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 3 (6) | 2 (2) | 3 (3) | 0 (0)
Folate deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral microhaemorrhage (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 3 (3) | 1 (1)
Cognitive disorder (Nervous system disorders) | 1 (1) | 2 (3) | 2 (2) | 3 (3) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 3 (4) | 2 (2) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Vasogenic cerebral oedema (Nervous system disorders) | 2 (2) | 2 (2) | 5 (5) | 3 (3) | 0 (0)
Aggression (Psychiatric disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Delusion (Psychiatric disorders) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Bapineuzumab program was discontinued prematurely. Efficacy results obtained after Week 78 are not presented due to the very small number of participants after this time point.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.